CLINICAL TRIAL: NCT04464798
Title: A Phase 1/2, Multicenter, Open-label Study to Assess Safety, Pharmacokinetics, and Preliminary Efficacy of CC-220, Alone and in Combination With an Anti-CD20 Monoclonal Antibody (mAb) in Subjects With Relapsed or Refractory Lymphomas.
Brief Title: A Dose Finding and Safety Study of CC-220, Alone and in Combination With an Anti-CD20 Monoclonal Antibody (mAb) in Subjects With Relapsed or Refractory Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-NHL-001; U1111-1254-1772 (Registry Identifier: WHO); 2020-000354-10 (EudraCT Number)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
Keywords: Relapsed or Refractory Lymphomas; Lymphomas; CC-220; Anti-CD20; Monoclonal Antibody; Pharmacokinetics; Safety
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — iberdomide; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A- Monotherapy in R/R lymphoma subjects (Experimental): Subjects with Relapsed or Refractory (R/R) lymphoma who have been allocated to Cohort A will receive CC-220 monotherapy (MonoT). Oral CC-220 at dose specified by cohort dose level from Day 1 to 21 of each 28-day cycle, up to PD or a maximum of 24 cycles.
  Interventions: Drug: CC-220
- Cohort B- CC-220 and rituximab in R/R B-Cell NHL subjects (Experimental): Subjects with R/R B-cell Non Hodgkin Lymphoma (NHL) who have been allocated to Cohort B will receive CC-220 in combination with rituximab.
  * Oral CC-220 at dose specified by cohort dose level from Day 1 to 21 of each 28-day cycle up to PD or maximum 24 cycles.
  * Rituximab will be administered at 375 mg/m2 IV at C1D1 and then on D8, D15, and D22 of C1 and then every 28-day cycle at D1 from C2 to C5, either by SC administration at a dose of 1400 mg or by IV infusion at a dose of 375 mg/m2.
  Interventions: Drug: CC-220; Drug: Rituximab
- Cohort C - CC-220 and obinutuzumab in R/R FL or MZL subjects (Experimental): Subjects with R/R FL (Grade 1 to 3a) or MZL who have been allocated to Cohort C will receive CC-220 in combination with obinutuzumab.
  * Oral CC-220 at dose specified by cohort dose level from Day 1 to 21 of each 28-day cycle, up to PD or a maximum of 12 cycles.
  * Obinutuzumab will be administered at 1000 mg at C1D1, D8, and D15, and on D1 of every 28-day cycle from C2 to C6.
  Interventions: Drug: CC-220; Drug: Obinutuzumab
- Cohort D -CC-220 monotherapy in participants with aggressive B-cell lymphoma and follicular lymphoma (Experimental)
  Interventions: Drug: CC-220
- Cohort E - CC-220 and rituximab in participants with aggressive B-cell lymphoma (Experimental)
  Interventions: Drug: CC-220; Drug: Rituximab
- Cohort F - CC-220 and rituximab with follicular lymphoma grade 1-3a (Experimental)
  Interventions: Drug: CC-220; Drug: Rituximab
- Cohort G - CC-220 plus obinutuzumab in participants with follicular lymphoma grade 1-3a (Experimental)
  Interventions: Drug: CC-220; Drug: Obinutuzumab

INTERVENTIONS:
Drug: CC-220 — Oral
  Other Names: Iberdomide
Drug: Rituximab — SC and IV infusion
  Arms: Cohort B- CC-220 and rituximab in R/R B-Cell NHL subjects; Cohort E - CC-220 and rituximab in participants with aggressive B-cell lymphoma; Cohort F - CC-220 and rituximab with follicular lymphoma grade 1-3a
Drug: Obinutuzumab — IV Infusion
  Arms: Cohort C - CC-220 and obinutuzumab in R/R FL or MZL subjects; Cohort G - CC-220 plus obinutuzumab in participants with follicular lymphoma grade 1-3a

SUMMARY:
This Phase 1/2, multicenter, open-label study to evaluate CC-220 alone, as well as in combination with an anti-CD20 mAb (rituximab or obinutuzumab) in subjects with relapsed or refractory (R/R) lymphoma. Subjects must have received at least 2 prior lines of therapy, and have at least one measurable lesion according to Lugano 2014 classification.

Study will consist of two parts: Part 1 (Dose Escalation) which will be followed by Part 2 (Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Has histologically confirmed (per local evaluation) diagnosis of lymphoma according to 2016 World Health Organization (WHO) classification including:

   1. Cohort A: all subtypes including B-cell, T-cell and Natural killer (NK)-cell Non-Hodgkin lymphoma (NHL), and Classical Hodgkin lymphoma (cHL).
   2. Cohort B: all B-cell NHL.
   3. Cohort C: FL Grade 1-3a and MZL including extranodal marginal zone lymphoma (ENMZL) of mucosa-associated lymphoid tissue (MALT lymphoma), nodal marginal zone lymphoma (NMZL) and splenic marginal zone lymphoma (SMZL)
   4. Cohort D: aggressive B-cell lymphoma and FL grade 1-3a
   5. Cohort E: aggressive B-cell lymphoma including DLBCL NOS, high-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements, Grade 3b FL and PMBCL
   6. Cohorts F and G: FL Grade 1 to 3a
3. Relapsed or refractory disease according to the following definitions:

   1. Aggressive B-cell lymphoma
   2. Follicular lymphoma (FL) and Marginal zone lymphoma (MZL): following at least 2 prior lines of systemic therapy (being previously exposed to at least 1 anti-CD20 mAb and 1 alkylating agent).
   3. Mantle cell lymphoma (MCL): following at least 2 prior lines of therapy including at least 1 immunochemotherapy and 1 bruton tyrosine kinase (BTK) inhibitor.
   4. Peripheral T-cell lymphoma (PTCL): following at least 2 prior lines of therapy OR after 1 prior line of standard therapy and being not eligible for any other approved regimen.
   5. Classical Hodgkin lymphoma (cHL): following at least 2 prior systemic lines of therapy and previously exposed to brentuximab vedotin and anti-PD1.
   6. All other subtypes: following at least 2 prior lines of therapy.
   7. Subjects previously treated with CAR-T therapy can be enrolled (irrespective of the indication).
4. Subjects must not be eligible for any other approved treatment for their underlying lymphoma as assessed by the Investigator.
5. Must have measurable disease defined by at least 1 fluorodeoxyglucose (FDG)-avid lesion for FDG-avid subtype and 1 bi-dimensionally measurable (> 1.5 cm in longest diameter) disease by computed tomography (CT) or magnetic resonance imaging (MRI), as defined by the Lugano classification. Site of measurable disease cannot be previously irradiated.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
7. Must have the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L or ≥ 1.0 x 109/L
   2. Hemoglobin (Hb) ≥ 8 g/dL.
   3. Platelets (Plt) ≥ 75 x 109/L or ≥ 50 x 109/L
   4. Aspartate aminotransferase / serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase / serum glutamic pyruvic transaminase (ALT/SGPT) ≤ 2.5 x ULN.
   5. Serum total bilirubin ≤ 1.5 ULN except in cases of Gilbert's syndrome, then ≤ 3.0 ULN.
   6. Estimated serum creatinine clearance of ≥ 50 mL/min
8. All subjects must:

   1. Have an understanding that the study drug could have a potential teratogenic risk.
   2. Agree to follow all requirements defined in the Pregnancy Prevention Program for CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
9. Females of childbearing potential (FCBP1) must:

   a. Have 2 negative pregnancy tests as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment.
10. Male subjects must:

    1. Practice true abstinence2 or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study,

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Any significant medical condition, active infection (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2) suspected or confirmed, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Life expectancy ≤ 3 months.
4. Diagnosis of lymphoblastic lymphoma.
5. Aggressive lymphoma relapse requiring immediate cytoreductive therapy to avoid potential life-threatening consequences (eg, due to tumor location).
6. Prior Grade 3 or 4 infusion related reaction with rituximab (for Cohorts B, E and F) or obinutuzumab (for Cohorts C and G).
7. Prior therapy with the cereblon-modulating drug CC-99282.
8. Chronic systemic immunosuppressive therapy or corticosteroids.
9. Prior ASCT ≤ 3 months prior to starting CC-220 or > 3 months AND with unresolved, Grade > 1, treatment-related toxicity.
10. Prior allogeneic stem cell transplant with either standard or reduced intensity conditioning ≤ 6 months prior to starting CC-220 or > 6 months with unresolved, Grade > 1, treatment-related toxicity.
11. Hypersensitivity to the active substance or to murine proteins, or to any of the other excipients of rituximab or obinutuzumab.
12. Known allergy to thalidomide, pomalidomide or lenalidomide.
13. Inability or unwilling to undergo protocol required thromboembolism prophylaxis.
14. Major surgery ≤ 2 weeks prior to starting CC-220;
15. Peripheral neuropathy ≥ Grade 2 (NCI CTCAE v5.0).
16. Documented or suspected central nervous system (CNS) involvement of disease.
17. Subject with clinically significant cardiac disease.
18. Known seropositivity for or active viral infection with human immunodeficiency virus (HIV).
19. Known chronic active hepatitis B
20. History of other malignancy, unless the subject has been free of the disease for ≥ 3 years; exceptions to the ≥ 3-year time limit include history of the following:

    1. Incidental histologic finding of prostate cancer (or prostate cancer that has been treated with curative intent

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | During the First cycle (each cycle is 28 days)
  is defined as the dose that satisfies the escalation with overdose control (EWOC) criterion that the posterior probability to have excessive toxicity is less than 25% and has the highest probability of dose-limiting toxicity (DLT) rate being in the target interval (0.16 to 0.33)
Recommended Phase 2 Dose (RP2D) | During the first Cycle (each cycle is 28 days)
  is defined as the dose that will be selected for dose expansion based on PK/Pd and MTD

SECONDARY OUTCOMES:
Adverse Events (AEs) | From first dose to 28 days after last subject discontinues study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Pharmacokinetics - Cmax | At Cycle1 Day15 and Cycle2 Day15 (each cycle is 28 days)
  Maximum plasma concentration
Pharmacokinetics - Ctrough | At Cycle1 Day15 and Cycle2 Day15 (each cycle is 28 days)
  Observed plasma concentration at the end of the dosing interval
Pharmacokinetics - AUC(TAU) | At Cycle1 Day15 and Cycle2 Day15 (each cycle is 28 days)
  Area under the plasma concentration-time curve from time zero to tau, where tau is the dosing interval
Pharmacokinetics - tmax | At Cycle1 Day15 and Cycle2 Day15 (each cycle is 28 days)
  Time to maximum plasma concentration
Pharmacokinetics - CLT/F | At Cycle1 Day15 and Cycle2 Day15 (each cycle is 28 days)
  Apparent total plasma clearance
Best Overall Response Rate (ORR) | Approximately 5 years
  is defined as the proportion of subjects with best overall response as either CR or partial response (PR) before subsequent anti-lymphoma therapy
Complete Response Rate (CRR) | Approximately 5 years
  is defined as the proportion of subjects experiencing CR before receiving any subsequent anti-lymphoma therapy
Time to Response (TTR) | Approximately 5 years
  is defined as the time from enrollment dose date to the date of first documented response (≥ PR)
Duration of Response (DOR) | Approximately 5 years
  is defined as the time from first dose date to the date of first documented response (≥ PR)
Progression-free Survival (PFS) | Approximately 5 years
  is defined as the time from enrollment date to the first occurrence of disease progression or death from any cause
Overall Survival (OS) | Approximately 5 years
  is defined as the time from enrollment date to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (6):
  - Local Institution - 106, Phoenix, Arizona
  - Local Institution - 105, Lake Mary, Florida
  - Local Institution - 102, Rochester, Minnesota
  - Local Institution - 100, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Local Institution - 103, Nashville, Tennessee
- France (6):
  - Local Institution - 203, Créteil
  - Local Institution - 200, Lillie Cedex
  - Local Institution - 201, Montpellier
  - Local Institution - 202, Nantes
  - Local Institution - 204, Paris
  - Local Institution - 205, Pessac
- Germany (4):
  - Local Institution - 401, Berlin
  - Local Institution - 402, Leipzig
  - Local Institution - 403, Münster
  - Local Institution - 404, Würzburg
- Italy (4):
  - Local Institution - 300, Brescia
  - Local Institution - 303, Milan
  - Local Institution - 301, Pavia
  - Local Institution - 302, Verona
- South Korea (3):
  - Local Institution - 502, Seoul
  - Local Institution - 501, Seoul
  - Local Institution - 500, Seoul
- Taiwan (3):
  - Local Institution - 600, Niaosong District Kaohsiung City
  - Local Institution - 601, Taoyuan
  - Local Institution - 602, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com